CLINICAL TRIAL: NCT05091944
Title: An Interactive Web-based Decision Aid for Shared Decision Making: Birth Choice After Cesarean in Taiwan
Brief Title: An Interactive Web-based Birth Decision Aid for Shared Decision Making
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taipei University of Nursing and Health Sciences (Other)
Responsible Party: Principal Investigator, She Wen Chen, Assistant Professor, National Taipei University of Nursing and Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2021-02-003A
Record Dates: First submitted 2021-09-14; First posted 2021-10-25 (Actual); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Shared Decision Making; Vaginal Birth After Cesarean
Keywords: communication aids; web-based decision aids

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention (Experimental): usual care plus web-based birth decision aid
  Interventions: Device: web-based birth decision aid
- control (No Intervention): ususal care

INTERVENTIONS:
Device: web-based birth decision aid — Women in the intervention group receive both usual care and decision support (an interactive web-based birth decision aid). The innovative interactive web-based birth decision aid comprised five components: Component 1-a communication aid video involves 2 expert's talk about how to participate in SDM and prepare self with choice talk, option talk and decision talk(10 minutes )and practice communication skills with clinician(10 minutes); Component 2-overall of the function and features of birth decision aid. Component 3-introduce the benefits and risk of vaginal birth after cesarean; Component 4- the benefits and risk of elective repeat cesarean section; Component 5 -a quit to confirm women's knowledge regarding the two choices and confirm women's values.
  Arms: intervention

SUMMARY:
An interactive web-based decision aid for shared decision making: birth choice after cesarean in Taiwan

Background: Taiwan has a high national caesarean rate coupled with a low vaginal birth after caesarean (VBAC) rate. Studies suggest that pregnant women do not receive sufficient information about birth choices after caesarean in Taiwan and shared decision making (SDM) is not an expectation. Chen conducted a pilot study. Improvements in knowledge for the decision aid group were larger than for the usual care group, although differences between groups were not statistically significant. An interactive multimedia technology and humanity communication may provide opportunities to increase engagement and support women during decision consultations. Following previous pilot study, the study aims to examine the effectiveness of an interactive web-based birth decision aid for SDM in pregnant women who have had a previous cesarean.

Methods: A quantitative approach will be conducted with a randomized pre-test and post-test experimental design in a medical center in northern Taiwan. Participants who have had one previous CS will be recruited at 14-16 weeks. A total of 172 women will be completed a baseline survey and will be randomly allocated to either the intervention (usual care plus an interactive web-based birth decision aid ) or usual care (general maternal health booklet) group. A follow up survey at 35-38 weeks measured change in decisional conflict, knowledge, birth preference and decision aid acceptability. Actual birth outcomes and satisfaction will be assessed one month after birth.

Contributions/ Implementation of clinical practice The study will potentially increase women and obstetricians to support VBAC and SDM. The interactive decision aid tool may reduce time-consumption for health education. Linking web-based data analysis of AI into medical record can be beneficial for clinical practice and research in the future.

DETAILED DESCRIPTION:
Study design:

A sequential mixed methods approach was conducted based on the Ottawa Decision Support Framework (ODSF). The current study will represent Aim 4 (Intervention implementation phase), comprising two stages. Stage 1 involves a randomized pre-test and post-test experimental design. Decisional conflict, knowledge, birth preference, and decision aid acceptability are assessed. Stage 2 consists of a survey, actual birth outcome and satisfaction are assessed.

Setting and participants:

The study will be conducted in a medical center in northern Taiwan. The medical center offers 24-hour system of the designated obstetrician. Using purposive sampling, the selection criteria include women who are medically eligible for VBAC in the study site, had experienced one previous CS, 14-16 weeks' gestation, had at least a half year interval between current pregnancy and the previous birth and are fluent in English or Mandarin. Exclusion criteria included women with multiple pregnancy, previous classic CS or myomectomy, and/or pregnancy with high risk of complications (for example, women who had risk factors such as hypertension, heart disease, diabetes, epilepsy, threatened premature labor, or another pre-existing medical problem).

Randomization:

Prior to the study commencing, the research team will conduct online discussions to clarify the research protocol. Eligible participants will be provided information about the study by the principal researcher and signed a written consent. Using computer permuted block randomization, participants will be allocated to control group (usual care) and intervention group (usual care plus the interactive web-based birth decision aid). After administering the baseline questionnaire, women will be allocated to the intervention group and give instructions by the principal researcher on how to log in the interactive birth decision aid platform/App. All participants confirm preferred mode of birth with their obstetrician prior to completing the second questionnaire.

Usual care:

A maternal health booklet, produced by Health Promotion Administration, Ministry of Health and Welfare, Executive Yuan, Taiwan, will be provided to all women. The booklet consists of 58 pages, presenting 5 "Dos" and 5 "Don'ts" during pregnancy. 5 "Dos" content included (1) Do receive prenatal exams according to schedule; (2) Do take good care during pregnancy; (3) Do recognize pregnancy complications; (4) Do know the signs of premature birth; (5) Do know the signs of labor. 5 "Don'ts" content included (1) Do not smoke or drink; (2) Do not be exposed to secondhand smoke; (3) Do not take medication without doctor's orders; (4) Do not choose a C-section in order to pick the time of birth; (5) Do not use drugs (52). There is very limited information relevant to mode of birth choice after caesarean.

Intervention:

Women in the intervention group will receive both usual care and decision support (an interactive web-based birth decision aid ). The interactive web-based birth decision aid will be modified from Professor Allison Shorten (English audio). We add communication aid at the beginning of platform/App. The communication aid comprises two components: components 1-how to participate in SDM and apply three talk to work together with clinicians (10 minutes) ; component 2-practice communication skill (10 minutes). Women will be assisted to create a unique username and password for secure decision aid access and its features and functions will be demonstrated. Intervention women will be invited to access the decision aid at home. All women are allowed to have many opportunities to access and use the decision aid during their pregnancy and will be recorded. They are encouraged to use the decision aid during recruitment and gestation visit in the Outpatient Department of Obstetrics. The principal researcher will provide 2-3 online consultations for individual women.

Outcome measures :

There are three primary and two secondary outcome measures. Primary outcome measures are decisional conflict, knowledge, birth preference and decision aid acceptability. Decisional conflict score (DCS)includes 16 questions in 5 sub-scale. Using the 5-point Likert 5 rating, from "strongly agree" ( 0 points) to "strongly disagree" (4 points). Knowledge measurement consists of a 15-item questionnaire asking participants to answer ''true,'' ''false,'' or ''unsure'' to a series of statements regarding risks and benefits of each birth mode. Previously tested Cronbach α for this questionnaire was = 0.67.

Secondary outcome measures are actual birth outcome and satisfaction. Satisfaction with decision scale (SWD) included six questions to measure women's satisfaction with their decision, using the Likert 5 rating, from "strongly agree" (5 points) to "strongly disagree" (1 points). Women have higher scores indicating increased SWD. Cronbach's α previously tested was 0.88.

Sample size :

Using G-POWER 3.1.9.2 software, sample size was calculated. Based on estimates from a previous pilot study, effect size=.40, a total of sample size 156 provides α = .05 and power = .80. To allow for preterm deliveries, mal-presentations, and losses to follow-up, an increase in the desired number by 10 percent would be 172.

Data collection and procedures :

Eligible women will be invited to participate in the study when they attend prenatal examination at the 14-16 weeks' gestation visit in the Outpatient Department of Obstetrics and Gynecology. After participants sign written consent for participation, women will be allocated to either the intervention group or control group. All participants will complete "personal basic information", "decision conflict scale" and "knowledge scale" in a quiet room. After completion of questionnaires, an interactive birth decision aid platform/App will be provided for intervention group women to discuss with their families at home. Individual consultations will be provided for intervention group women, by the principal researcher, at least twice during the 17-34 weeks' gestation period. All participants will complete "decision conflict scale" and "knowledge scale" and "decision aid acceptability at 35-38 weeks' gestation. A follow-up is held one month after birth. Postnatal women will be asked about "actual birth outcomes '' and complete a "satisfaction" questionnaire when they attend their postnatal examination visit .

Data analysis:

Quantitative data is managed and analyze using IBM SPSS Version 26.0. In terms of DCS and knowledge scores, matched pairs t-tests are used to compare differences between groups in change between pre and post test scores.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women had experienced one previous cesarean
* pregnant women had at least a half year interval between current pregnancy and the previous birth

Exclusion Criteria:

* women are multiple pregnancy
* women had previous classic CS or myomectomy
* pregnant women have high risk of complications

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — pregnant women
Enrollment: 86 (Estimated)
Dates: Start 2021-09-15 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
change is being assessed-decisional conflict | 14-16 week gestation and 35-38week gestation
  Decisional conflict score (DCS)includes 16 questions. Using the 5-point Likert 5 rating, from "strongly agree" (0 points) to "strongly disagree" (4 points)
change is being assessed-knowledge | 14-16 week gestation and 35-38week gestation
  Knowledge measurement consists of a 15-item questionnaire asking participants to answer ''true,'' ''false,'' or ''unsure'' to a series of statements regarding risks and benefits of each birth mode
change is being assessed-birth preference | 14-16 week gestation and 35-38week gestation
  VBAC/ERCS
decision aid acceptability | 35-38week gestation
  Decision aid acceptability included nine questions to measure women's acceptability regarding decision aid , using the Likert 5 rating, from "not at all" (1 points) to "a great deal" (5 points)

SECONDARY OUTCOMES:
Actual birth outcomes | one month after birth
  VBAC or ERCS
satisfaction of decision | one month after birth
  Satisfaction with decision scale (SWD) included six questions to measure women's satisfaction with their decision, using the Likert 5 rating, from "strongly agree" (5 points) to "strongly disagree" (1 points).

CONTACTS AND LOCATIONS:
Overall Officials: Shu Wen Chen, PhD, Principal Investigator — National Taipei University of Nursing and Health Science
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Chen SW, Shorten A, Yeh CC, Kao CH, Lu YY, Hu HW. An innovative web-based decision-aid about birth after cesarean for shared decision making in Taiwan: study protocol for a randomized control trial. Trials. 2023 Feb 9;24(1):103. doi: 10.1186/s13063-023-07103-8. PMID 36759893